CLINICAL TRIAL: NCT03213132
Title: An Insomnia Internet Intervention for Older Adults
Brief Title: Sleep Healthy Using The Internet for Older Adult Sufferers of Insomnia and Sleeplessness
Acronym: SHUTiOASIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Laval University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Karen Ingersoll, Professor, Department of Psychiatry and Neurobehavoiral Sciences, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-0089-00; R01AG047885 (NIH)
Record Dates: First submitted 2017-07-03; First posted 2017-07-11 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Insomnia; Sleep Initiation and Maintenance Disorders
Keywords: sleep; insomnia; CBT
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHUTi for older adults (Experimental): Participants will be assigned to the SHUTi (Sleep Healthy Using the Internet) online intervention optimized for older adults. They will spend 1-2 hours each week for 6-9 weeks completing daily sleep diaries as well as interactive core content covering topics of sleep behaviors, sleep thoughts, sleep education, and relapse prevention targeting issues specific to older adults. As users progress through the intervention, they will receive automated, tailored instructions for how to improve their sleep.
  Interventions: Behavioral: SHUTi (Sleep Health Using the Internet)
- SHUTi for older adults with stepped care (Active Comparator): Participants will be assigned to the SHUTi (Sleep Healthy Using the Internet) online intervention optimized for older adults. This is the same intervention as the first arm but with the addition of personalized emails or phone calls to participants by study personnel at specific time points as a result of not completing assigned tasks.
  Interventions: Behavioral: SHUTi (Sleep Health Using the Internet)
- Patient Education website (Placebo Comparator): Participants will be assigned to a relevant patient education website. It will include information about insomnia symptoms, diagnosis, prognosis, and information about CBT strategies for the older adult. Unlike SHUTi, the content will not be tailored and will be presented all at once.
  Interventions: Behavioral: Patient Education

INTERVENTIONS:
Behavioral: SHUTi (Sleep Health Using the Internet) — Cognitive Behavioral Therapy for insomnia delivered online and metered out over 6 weeks in a fully automated, interactive, tailored web-based program
  Other Names: CBTi
  Arms: SHUTi for older adults; SHUTi for older adults with stepped care
Behavioral: Patient Education — Educational website containing information on insomnia
  Other Names: Information
  Arms: Patient Education website

SUMMARY:
This study will compare the efficacy of an interactive internet intervention for older adults with insomnia called SHUTi OASIS (Sleep Healthy Using the Internet for Older Adult Sufferers of Insomnia and Sleeplessness) accessed at www.shutioasis.org both with and without support for adherence to that of a static educational website to improve sleep, health, mood, and overall quality of life.

DETAILED DESCRIPTION:
Insomnia is a significant public health problem for older adults with substantial medical, psychological and financial ramifications. With as many as 20-30% of older adults (age ≥55) meeting diagnostic criteria for chronic insomnia, finding accessible, effective, and low-cost treatments is critical. Cognitive-Behavioral Therapy for Insomnia (CBT-I) is a non-pharmacological intervention that has been shown to be efficacious when tailored for older adults. Regrettably, access to this treatment is significantly limited by a lack of trained clinicians and expense. To overcome barriers to face-to-face care, use of the Internet has emerged as a feasible and effective method to provide health information and treatment. Unfortunately, the health care field has been reluctant to use technology-delivered solutions with older patients out of a concern that older adults either do not have access to or do not want to use technology. However, older adults in the U.S. are the largest growing group of Internet users, and they generally have a desire to learn new technologies. When older adults do use technology-based programs for health promotion, they rate these programs favorably. Internet-delivered CBT-I for older adults has a high likelihood of major public health impact by allowing widespread access to a needed intervention, increasing the convenience of obtaining care, and decreasing treatment costs among an age group with high rates of insomnia known to exacerbate other concerns (health, mood, cognition).

The SHUTi Program: SHUTi is a self-guided (i.e., automated), interactive, and tailored web-based program modeled on the primary tenants of face-to-face CBT-I (sleep restriction, stimulus control, cognitive restructuring, sleep hygiene, relapse prevention). Intervention content is metered out over time through 6 "Cores." Users obtain access to a new Core based on a time and event-based schedule (e.g., 7 days after completion of previous Core). This schedule is consistent with the recommendation from a task force commissioned by the Academy of Sleep Medicine, which deemed that an average of 6 - 8 sessions constitutes "adequate treatment exposure". The SHUTi program relies on user-entered online Sleep Diaries to track progress and to tailor treatment recommendations (i.e., assign a "sleep restriction" window). Each Core acts as an online analog for the weekly sessions typically used when delivering CBT-I in a face-to-face format, following the same general structure: 1) Core objectives (what will be learned and why this information is important), 2) review of previous week's homework and sleep diary data, 3) new intervention material, 4) assignment of homework (treatment strategies for the coming week), and 5) a summary of the Core's main points. Intervention content is enhanced through a variety of interactive features, including personalized goal-setting, graphical feedback based on inputted symptoms, animations / illustrations to enhance comprehension, quizzes to test user knowledge, patient vignettes, and video-based expert explanation. Automated emails are also sent to encourage program adherence.

Participants in this study will be randomly assigned for a period of 9 weeks to one of three conditions: (1) the online CBT-i intervention optimized for older adults (SHUTi), (2) the online CBT-i intervention optimized for older adults (SHUTi) with additional adherence and technical support provided (stepped care), or (3) the patient education website. All participants will complete questionnaires and two weeks of daily sleep diaries about their symptoms at four time points - at the beginning of the study (baseline), immediately after completing the 9 week intervention (post), and at 6 and 12 months later.

ELIGIBILITY:
Inclusion Criteria:

* age 55 and over
* sleep onset latency (SOL) and/or wake after sleep onset (WASO) (>30 minutes for at least 3 nights/week)
* insomnia symptoms for ≥ 3 months
* no more than 6.5 hours of sleep per night
* the sleep disturbance (or associated daytime fatigue) must cause significant distress or - impairment in social, occupational, or other areas of functioning
* regular access (at least 2/week) and willingness to use a computer and the Internet and check email
* ability to read and speak English
* resident of the US

Exclusion Criteria:

* irregular sleep schedules that prevent the ability to follow intervention recommendations(i.e., with usual bedtimes outside of 8:00pm to 2:00am or arising time outside of 4:00am to 10:00am)
* current psychological treatment for insomnia
* initiated psychological or psychiatric treatment within past 3 months
* screen positive for a history of psychotic or bipolar disorder; and current severe depression, high risk of suicide, substance use (alcohol, drug) disorder within the past year
* symptoms suggestive of untreated sleep disorders other than insomnia (e.g., obstructive sleep apnea, restless legs syndrome, periodic limb movement disorder)
* presence of severe cognitive impairment
* presence of uncontrolled medical condition that is deemed to interfere with the study procedures, or put the study participant at undue risk

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Primary Sleep Outcome: Change in overall insomnia severity | Baseline, 9 weeks, 6 months, 1 year
  Insomnia Severity Index (ISI)

SECONDARY OUTCOMES:
Sleep variables: Change in wake after sleep onset (WASO) | Baseline, 9 weeks, 6 months, 1 year
  Consensus sleep diary questions
Sleep variables: Change in sleep onset latency (SOL) | Baseline, 9 weeks, 6 months, 1 year
  Consensus sleep diary questions
Daytime variables: change in attention and concentration | Baseline, 9 weeks, 6 months, 1 year
  Multiple Ability Self-Report Questionnaire
Daytime variables: change in levels of fatigue | Baseline, 9 weeks, 6 months, 1 year
  Fatigue Symptom Inventory
Daytime variables: change in mood (levels of depression and anxiety) | Baseline, 9 weeks, 6 months, 1 year
  Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Karen Ingersoll, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ritterband LM, Thorndike FP, Ingersoll KS, Lord HR, Gonder-Frederick L, Frederick C, Quigg MS, Cohn WF, Morin CM. Effect of a Web-Based Cognitive Behavior Therapy for Insomnia Intervention With 1-Year Follow-up: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Jan 1;74(1):68-75. doi: 10.1001/jamapsychiatry.2016.3249. PMID 27902836
- [Background] Morin CM, Bootzin RR, Buysse DJ, Edinger JD, Espie CA, Lichstein KL. Psychological and behavioral treatment of insomnia:update of the recent evidence (1998-2004). Sleep. 2006 Nov;29(11):1398-414. doi: 10.1093/sleep/29.11.1398. PMID 17162986
- [Background] Ritterband LM, Thorndike FP, Gonder-Frederick LA, Magee JC, Bailey ET, Saylor DK, Morin CM. Efficacy of an Internet-based behavioral intervention for adults with insomnia. Arch Gen Psychiatry. 2009 Jul;66(7):692-8. doi: 10.1001/archgenpsychiatry.2009.66. PMID 19581560
- [Derived] Shaffer KM, Daniel KE, Frederick C, Buysse DJ, Morin CM, Ritterband LM. Online sleep diaries: considerations for system development and recommendations for data management. Sleep. 2023 Oct 11;46(10):zsad199. doi: 10.1093/sleep/zsad199. PMID 37480840
- See also: Center for Behavioral Health and Technology at the University of Virginia — http://bht.virginia.edu